CLINICAL TRIAL: NCT03359382
Title: The Rehabilitation Effect of Exercise Training in Cruciate Ligament Reconstruction Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wei-Hsiu Hsu, PI, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CORPG6G0271-3
Record Dates: First submitted 2017-11-19; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: ACL Injury; ACL - Anterior Cruciate Ligament Rupture; ACL - Anterior Cruciate Ligament Deficiency
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention)
- exercise (Experimental)
  Interventions: Other: Resistance or home exercise combined with eccentric exercise

INTERVENTIONS:
Other: Resistance or home exercise combined with eccentric exercise — First year: Progressive resistance exercise (60-80% RM) combined with low intensity eccentric exercise (10%RM).
  Second year: Progressive resistance exercise (60-80% RM) combined with progressive eccentric exercise (10-80% RM).
  Third year:Home exercise combined with low intensity eccentric exercise (10% RM )
  Arms: exercise

SUMMARY:
After anterior cruciate ligament (ACL) injury, the involved quadriceps may demonstrate weakness due to decrease in quadriceps activation. However, elapsed time from the injury may affect muscle strength by restoration of the quadriceps activation. The injury is characterized by joint instability that leads to decreased activity, unsatisfactory knee function, and poor knee-related quality of life in the short term, and it is associated with an increased risk of osteoarthritis on the knee. This study was designed to compare muscle strength, questionnaire and knee function in patients with different exercise training.

ELIGIBILITY:
Inclusion Criteria:

* cruciate ligament rupture patients

Exclusion Criteria:

* Central nervous or peripheral neuropathy, or those with cardiovascular disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from preoperative muscle mass | One day after rupture of the cruciate ligament, one day before operative, postoperative 4 months, 7 months, 12 months, 24 months
  Muscle mass measurement is measured by dual-energy x-ray absorptiometry (DXA). DXA measures the muscle mass of the whole body

SECONDARY OUTCOMES:
Change from preoperative motion analysis | One day after rupture of the cruciate ligament, one day before operative, postoperative 4 months, 7 months, 12 months, 24 months
  An optoelectronic eight-camera Vicon motion analysis system (T20; Oxford Metrics Ltd., Oxford, United Kingdom) was used to capture three dimensional (3D) kinematic data at 100 Hz during five walking trials. Two force plates (OR6, AMTI, Watertown, Massachusetts) embedded in the floor were synchronised with the motion capture system to record ground reaction force (GRF) during walking at a sampling rate of 1000 Hz.
Change from preoperative muscle strength | One day after rupture of the cruciate ligament, one day before operative, postoperative 4 months, 7 months, 12 months, 24 months
  The muscle strength of the lower extremity including hip flexor/extensor, knee flexor/extensor, and ankle plantar flexor/dorsiflexor were tested by HUMAC NORM system (CSMi, U.S.A.) with the mode of concentric/concentric contraction at the angular velocity of 60 degree/s.
Change from preoperative body composition questionnaire assessment | One day after rupture of the cruciate ligament, one day before operative, postoperative 4 months, 7 months, 12 months, 24 months
  Body composition was assessed using an eight-polar tactile-electrode impedance meter (InBody 720; Biospace, Seoul, Korea), which simultaneously recorded bodyweight, total body fat mass, total body muscle mass, lean body mass, bone mineral content and basal metabolic rate.
Change from preoperative surface electromyography | One day after rupture of the cruciate ligament, one day before operative, postoperative 4 months, 7 months, 12 months, 24 months
  Quadriceps and hamstrings EMG amplitudes were assessed during walking with stand phase using surface electromyography (EMG) sampled at 1000 Hz (BioNomadix, BIOPAC systems, Inc, Goleta, CA) with electrodes placed over the vastus medialis (VM), vastus lateralis (VL), rectus femoris (RF) and biceps femoris (BF).
Change from preoperative hop test | One day after rupture of the cruciate ligament, one day before operative, postoperative 4 months, 7 months, 12 months, 24 months
  Include: single leg vertical hop, Single leg forward one-step hop, Single leg three-step hop, single leg three-step crossover hop. Record hop height, distance and completion of action time.
Change from preoperative fitness | One day after rupture of the cruciate ligament, one day before operative, postoperative 4 months, 7 months, 12 months, 24 months
  Fitness of all subjects was evaluated using the HELMAS Physical Fitness Management System (Seoul, Korea). Several dimensions of health-related fitness were evaluated, including muscular strength (grip strength and back strength); balance (closed-eye foot balance); cardiorespiratory endurance (step test); flexibility (sitting trunk flexion and trunk extension); muscle endurance (sit-ups); and agility (reaction time and side steps).
Marx activity rating scales questionnaire assessment | one day before operative
  The Marx activity rating scales is a patient-reported instrument. Contrary to the construction of activity level in the Tegner, which is based on participation in specific work and sports activities, activity level of the Marx is determined by measuring some components of physical function that are common to the most sporting activities.
Change from preoperative SF-36 questionnaire assessment | One day after rupture of the cruciate ligament, one day before operative, postoperative 4 months, 7 months, 12 months, 24 months
  SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower score the more disability. The higher the score the less disability. Eight sections including physical function, role limitation due to physical problems, bodily pain, general health, vitality, social functioning, role limitation due to emotional problems, and mental health. Additionally, the eight health domains can be used to provide a physical component summary and mental component summary score.
Change from preoperative KOOS questionnaire assessment | One day after rupture of the cruciate ligament, one day before operative, postoperative 4 months, 7 months, 12 months, 24 months
  KOOS contains 5 subscales with a total of 42 items: 1) pain, 2) other symptoms, 3) function in daily living (ADL), 4) function in sport and recreation and 5) knee-related quality of life. Each question receives a score from 0 to 4 and the scores are transformed to a 0-100 score (0, extreme symptoms, 100, no symptoms). The User's Guide, is available from www.koos.nu.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Hsiu Hsu, Dr., Study Chair — Sports Medicine Center, Chang Gung Memorial Hospital at Chia Yi, Chia Yi, Taiwan
Locations (1):
- Sports Medicine Center, Chang Gung Memorial Hospital, Chiayi City, Taiwan